CLINICAL TRIAL: NCT03000166
Title: Step-Up Intervention for Self-Management of Fatigue in Young Adults Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Froedtert Hospital (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jeanne M. Erickson, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P20NR015339-PP3; P20NR015339 (NIH)
Record Dates: First submitted 2016-12-15; First posted 2016-12-21 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Young Adult, Cancer, Physical Activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step-Up Intervention Group (Experimental): Participants assigned to the Step-up intervention group will receive a 12-week physical activity intervention which includes components of education, negotiated collaboration to set individual physical activity goals during chemotherapy cycles, and tools for self-monitoring of physical activity.
  Interventions: Behavioral: Step-Up Intervention
- Attention Control Group (No Intervention): Participants assigned to the attention control group will receive usual guidance about maintaining physical activity during chemotherapy from their oncology providers.

INTERVENTIONS:
Behavioral: Step-Up Intervention — Intervention group participants will meet with a study facilitator during 5 regularly scheduled visits for chemotherapy. The facilitator will provide education about the benefits of physical activity and strategies to overcome barriers to physical activity, help the participants to set physical activity goals based on ability and preferences, and educate the participant on using a physical activity tracker.
  Arms: Step-Up Intervention Group

SUMMARY:
The purpose of the study is to determine the impact of a physical activity intervention on the self-management of fatigue in young adults receiving chemotherapy. Half of the participants will receive an intervention which includes education and resources to set physical activity goals and monitor progress toward goals.

DETAILED DESCRIPTION:
Interventions to increase physical activity have been shown to relieve fatigue in patients receiving chemotherapy, but no studies have tested a physical activity intervention to improve fatigue in young adults receiving chemotherapy. This study will determine the impact of a physical activity intervention on the self-management process variables of self-efficacy and self-regulation and their relationships to physical activity and fatigue severity in young adults receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of cancer;
* are within the first two months of a chemotherapy regimen that will last at least another 3 months;
* are ambulatory without assistance;
* have written consent from their physician to participate;
* have the ability to understand English;
* have access to a computer and the Internet.

Exclusion Criteria:

* symptoms of uncontrolled cardiopulmonary disease, neurological disease
* delayed wound healing
* high risk of bone fracture
* pre-existing peripheral neuropathy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Schiffman, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (2):
- United States (2):
  - Froedtert Hospital, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 471 screened participants, 67 met inclusion criteria and were invited to participate in the study. 47 agreed to participate. 25 were randomized to the Step-Up intervention group, and 22 were randomized to the attention control group.
Groups:
- Step-up Intervention Group: Participants assigned to the intervention group will receive a 12-week physical activity intervention which includes components of education, negotiated collaboration to set individual physical activity goals during chemotherapy cycles, and tools for self-monitoring of physical activity.
  Step-Up Intervention: Intervention group participants will meet with a study facilitator during 5 regularly scheduled visits for chemotherapy. The facilitator will provide education about the benefits of physical activity and strategies to overcome barriers to physical activity, help the participants to set physical activity goals based on ability and preferences, and educate the participant on using a physical activity tracker.
Period: Overall Study
Arm/Group | Step-up Intervention Group | Attention Control Group
Started | 25 | 22
Completed | 25 | 19
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Step-Up Intervention Group | Attention Control Group | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.96 (4.71) | 32.77 (5.79) | 32.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 5 | 25
  Male | 5 | 17 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 21 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Fatigue [Mean (Standard Deviation); unit: units on a scale] — PROMIS Fatigue Short form. Participants self-report their fatigue over the past 7 days using the 8-item PROMIS Fatigue Short Form. The response scale is a 5-point Likert scale (1-never to 5-always). Raw scores can range from 8-40. Raw scores are converted to standardized T-scores, with higher scores indicating greater fatigue severity. T-Scores range from 33.1 - 77.8. A T-score of 50 represents the average fatigue severity of a national sample of the general US population. A score over 50 represents a person with more than average fatigue while a score under 50 is less than average fatigue.
  units on a scale | 54.2 (10.6) | 56.6 (7.8) | 55.3 (9.4)
Light Intensity Physical Activity [Mean (Standard Deviation); unit: minutes/day] — As measured with a waist-worn accelerometer. The accelerometer counts the number of times a person moves forward in a certain time period (counts per minute). Accelerometer data was analyzed using the ActiLife software (v13.3). Freedson adult cutpoints in counts per minute (cpm) were applied to assess time spent in sedentary (0-99 cpm), light (100-2019 cpm), moderate (2020-5998 cpm), and vigorous (>5999 cpm) physical activity. The intensity of physical activity corresponds to the energy expended by that individual. Light intensity physical activity requires the least amount of effort.
  minutes/day | 228.7 (61.3) | 208.7 (60.1) | 220.27 (60.8)
Moderate intensity physical activity [Mean (Standard Deviation); unit: minutes/day] — As measured by waist-worn accelerometer. The accelerometer counts the number of times a person moves forward in a time points. Accelerometer data was analyzed using the ActiLife software. Freedson adult cutpoints in counts per minute (cpm) were applied to assess time spent in sedentary (0-99 cpm), light (100-2019 cpm), moderate (2020-5998 cpm), and vigorous (>5999 cpm) physical activity. The intensity of physical activity corresponds to the energy expended by that individual. Moderate intensity physical activity requires medium effort, such as walking fast.
  minutes/day | 13.2 (19.9) | 15.3 (20.0) | 14.1 (19.7)
Steps/day [Mean (Standard Deviation); unit: steps/day] — As measured by a waist-worn accelerometer. Steps per day were calculated using algorithms that were based on records of accelerations (forward movements) that occur during ambulation (walking). Around 10,000 steps/day is a reasonable number of steps recommended as activity for healthy adults.
  steps/day | 4227.4 (2429) | 4288.8 (2545) | 4253.2 (2444)
Self-efficacy for Physical Activity [Mean (Standard Deviation); unit: units on a scale] — As measured by the Physical Activity Assessment Inventory (PAAI).The PAAI is a 13-item scale and was developed to measure confidence to be physically active under various conditions. Responses are measured on a 100-point scale, ranging from 0 ("cannot do at all") to 100 ("certain can do"). An average score is calculated, and a higher score indicates greater self-efficacy. Higher scores that mean more confidence in the ability to be physically active in various conditions would be a positive outcome.
  units on a scale | 62.7 (23.4) | 59.4 (24.4) | 61.2 (4.2)
Self-regulation for Physical Activity [Mean (Standard Deviation); unit: units on a scale] — As measured by the Index of Self-Regulation (ISR).The ISR is a 9-item scale that measures levels of self-regulation, which includes ability to process information, monitor performance, and take action in relation to goals. Responses are measured on a 6-point Likert scale (1=strongly disagree to 6=strongly agree), and scores can range from 9-54. An average score is calculated, and a higher score indicates a higher level of self-regulation. Higher scores indicating a higher level of self-regulation is a positive outcome.
  units on a scale | 4.24 (1.10) | 4.10 (0.99) | 4.18 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Self-efficacy for Physical Activity
Description: Physical Activity Assessment Inventory (Haas & Northam, 2010) The scale measures confidence to be physically active under various conditions. Scores range from 0=cannot do at all to 100=certain can do.
Time Frame: Completion of post-study measures (average 15 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Step-Up Intervention Group | Attention Control Group
Number analyzed (Participants) | 25 | 19
score on a scale | 62.6 (22.9) | 56.2 (24.4)
Statistical Analysis 1: Comparison: Step-Up Intervention Group vs Attention Control Group; Test type: Superiority; p = 0.22, Mixed Models Analysis

2. Primary Outcome: Self-regulation of Physical Activity
Description: Index of Self-Regulation (Yeom et al., 2011) The scale measures self-regulation skills, including processing information, monitoring performance, and taking action to meet goals. Scores range from 1 to 6, with higher scores indicating agreement that the individual has these skills.
Time Frame: Completion of post-study measures (average 15 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Step-Up Intervention Group | Attention Control Group
Number analyzed (Participants) | 25 | 19
score on a scale | 4.7 (0.8) | 4.4 (1.1)
Statistical Analysis 1: Comparison: Step-Up Intervention Group vs Attention Control Group; Test type: Superiority; p = 0.40, Mixed Models Analysis

3. Secondary Outcome: Steps Per Day
Description: Measured by accelerometer
Time Frame: Completion of post-study measures (average 15 weeks)
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Step-up Intervention Group | Attention Control Group
Number analyzed (Participants) | 16 | 15
steps per day | 4720 (3772) | 3991 (2428)
Statistical Analysis 1: Comparison: Step-up Intervention Group vs Attention Control Group; Test type: Superiority; p = 0.17, Mixed Models Analysis

4. Secondary Outcome: Fatigue Severity
Description: Measured with PROMIS - Fatigue Short Form Fatigue severity is measured over the past 7 days from 1=never to 5=always. The raw scores are converted to T-scores, where 50=average fatigue in the general population. Higher scores indicate greater fatigue severity.
Time Frame: Completion of end-of-study measures (average 15 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Step-up Intervention Group | Attention Control Group
Number analyzed (Participants) | 25 | 19
score on a scale | 53.6 (7.2) | 57.4 (8.9)
Statistical Analysis 1: Comparison: Step-up Intervention Group vs Attention Control Group; Test type: Superiority; p = 0.20, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Data related to adverse events were collected over the duration of the time each participant was on study. Participants were considered on study from the date of enrollment through the completion of completion of post-study data collection. The average time for each participant to be on study was 15 weeks, but ranged from 10-23 weeks due to variations in the timing of their chemotherapy as well as completion of post-study measures.
Description: Adverse events were defined as serious or not serious.
Arm/Group | Step-up Intervention Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03000166/Prot_SAP_000.pdf